CLINICAL TRIAL: NCT05808478
Title: Augmentative Alternative Communication Intervention Delivered Via Eye-tracking Technology
Brief Title: Eye-tracking Technology for Severe Communication Disability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Francesca Cucinotta, Principal Investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EYETRACK01
Record Dates: First submitted 2023-03-17; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Communication Disabilities
Keywords: Augmentative and Alternative Communication, Eye tracker, Communication Disabilities
MeSH Terms: conditions — Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG) (Experimental): The experimental group will undergo treatment with innovative high-tech tools, such as Eye Tracking, for communication purposes. The duration of the treatment will be six months, twice a week, with sessions of 45 minutes.
  Interventions: Behavioral: AAC + Eye Tracking
- Control Group (CG) (Active Comparator): The control group will undergo conventional AAC treatment, with low-tech tools, such as PECS or sign language.
  The duration of the treatment will be six months, twice a week, with sessions of 45 minutes.
  Interventions: Behavioral: AAC

INTERVENTIONS:
Behavioral: AAC + Eye Tracking — The AAC treatment will be supported by the use of an innovative high-tech tool, such as Eye Tracking. The duration of treatment will be 6 months, with sessions of 45 minutes twice a week.
  Arms: Experimental Group (EG)
Behavioral: AAC — Treatment involves the use of conventional AAC, with low-tech tools, such as PECS or sign language. The duration of treatment will be six months, twice a week, with sessions of 45 minutes.
  Arms: Control Group (CG)

SUMMARY:
The aim of this project is to develop an Augmentative and Alternative Communication intervention through the use of Eye tracker system.

DETAILED DESCRIPTION:
The term "complex communication needs" includes all patients who present severe disturbances in speech and language production and/or in comprehension, in relation to oral or written communication modalities. The main purpose of Augmentative and Alternative Communication (AAC) is to promote the best possible communication for people with complex communication needs, through the use of techniques, methods and tools aimed not at replacing pre-existing communication methods but at increasing skills of natural communication through the enhancement of present skills. The Eye tracker system, thanks to allows the recording and analysis of eye movements, could be used successfully to support communication in patients with severe communication disability.

The goal of this study is to develop an efficacy Augmentative and Alternative Communication intervention using eye-tracking technology for patients with severe communication disability.

The secondary objective was to examine the psychosocial impact of technology for AAC on parents' perspectives and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* aged between 3 and 17 years affected by neuropsychiatric pathology presenting complex communication needs
* Control of eye motility and visual fixation
* ability to maintain position in front of the monitor
* availability of at least one member of the family nucleus to participate in the therapeutic process
* cognitive skills appropriate to the task such as being able to recognize images and being able to memorize procedures necessary to use the various basic functions

Exclusion Criteria:

* age not between 3 and 17 years
* difficulty in controlling ocular motility and visual fixation
* the unavailability of at least one member of the family nucleus to participate in the therapeutic process
* impaired cognitive skills on the task such as being able to recognize pictures and being able to memorize procedures necessary to use various basic functions

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-01-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MacArthur-Bates Communicative Development Inventory | Month 0
  The MacArthur-Bates Communicative Development Inventory is a questionnaire for parents. This is used for the study and evaluation of communication and language in children with typical and atypical development.
MacArthur-Bates Communicative Development Inventory | Month 3
  The MacArthur-Bates Communicative Development Inventory is a questionnaire for parents. This is used for the study and evaluation of communication and language in children with typical and atypical development.
MacArthur-Bates Communicative Development Inventory | Month 6
  The MacArthur-Bates Communicative Development Inventory is a questionnaire for parents. This is used for the study and evaluation of communication and language in children with typical and atypical development.
Communication Matrix | Month 0
  is an online assessment tool created to help professionals and family members support people with severe communication disorders on their journey to greater self-expression. Total score on an assessment of early expressive communication skills.
Communication Matrix | Month 3
  is an online assessment tool created to help professionals and family members support people with severe communication disorders on their journey to greater self-expression. Total score on an assessment of early expressive communication skills.
Communication Matrix | Month 6
  is an online assessment tool created to help professionals and family members support people with severe communication disorders on their journey to greater self-expression. Total score on an assessment of early expressive communication skills.
Interactive Check list for Augmentative Communication | Month 0
  Interactive Check list for Augmentative Communication is an observational tool for evaluating interactive behavior
Interactive Check list for Augmentative Communication | Month 3
  Interactive Check list for Augmentative Communication is an observational tool for evaluating interactive behavior
Interactive Check list for Augmentative Communication | Month 6
  Interactive Check list for Augmentative Communication is an observational tool for evaluating interactive behavior

SECONDARY OUTCOMES:
The World Health Organization Quality of Life | T0 (Baseline) - T1 (3 months) - T2 (6 months)
  The World Health Organization Quality of Life -BREF consists of 26 questions. The World Health Organization Quality of Life -BREF has Likert-type scoring ranging from 1 to 5. As the score obtained from the sub-domains of the scale increases, the quality of life increases.
Parenting Stress Index | T0 (Baseline) - T1 (3 months) - T2 (6 months)
  Measures parenting stress
Forerunners in Communication - ComFor | T0 (Baseline) - T1 (3 months) - T2 (6 months)
  Forerunners in Communication assesses the precursors of augmentative communication. It measures the ability to perceive and attribute meanings to forms of communication
Vineland Adaptive Behavior Scales II | T0 (Baseline) - T1 (3 months) - T2 (6 months)
  The Vineland Adaptive Behavior Scales are a standardized semi-structured interview to measure adaptive behavior, among the most sensitive to change in autism research. Standard scores have a mean of 100 and a standard deviation of 15.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neurolesi Bonino Pulejo, Messina, Italy

REFERENCES:
- [Background] Mirenda P, Eicher D, Beukelman DR. Synthetic and natural speech preferences of male and female listeners in four age groups. J Speech Hear Res. 1989 Mar;32(1):175-83. doi: 10.1044/jshr.3201.175. PMID 2523007
- [Background] Corallo F, Bonanno L, Lo Buono V, De Salvo S, Rifici C, Pollicino P, Allone C, Palmeri R, Todaro A, Alagna A, Bramanti A, Bramanti P, Marino S. Augmentative and Alternative Communication Effects on Quality of Life in Patients with Locked-in Syndrome and Their Caregivers. J Stroke Cerebrovasc Dis. 2017 Sep;26(9):1929-1933. doi: 10.1016/j.jstrokecerebrovasdis.2017.06.026. Epub 2017 Jul 18. PMID 28733123
- [Background] Uliano D, Falciglia G, Del Viscio C, Picelli A, Gandolfi M, Passarella A. Augmentative and alternative communication in adolescents with severe intellectual disability: a clinical experience. Eur J Phys Rehabil Med. 2010 Jun;46(2):147-52. Epub 2010 Apr 13. PMID 20485219